CLINICAL TRIAL: NCT04465461
Title: A Pilot Study of Video Assisted Thoracic Surgery (VATS) Fissure Completion Prior to Zephyr® Endobronchial Valve Insertion for Severe Chronic Obstructive Pulmonary Disease (COPD) in Patients With COllateral VEntilation
Brief Title: Video Assisted Thoracic Surgery (VATS) Fissure Completion Prior to Zephyr® Endobronchial Valve Insertion
Acronym: COVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulmonx Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 630-0026-01
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Emphysema
MeSH Terms: conditions — Pulmonary Emphysema | interventions — Thoracic Surgery, Video-Assisted; Pneumonectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): Patients exhibiting baseline collateral ventilation by Chartis® balloon catheter assessment who undergo video-assisted thoracoscopic surgery (VATS) fissure completion surgery, confirmation of fissure completion by computerized tomography (CT) scan and confirmation of conversion to collateral ventilation negative by Chartis® balloon catheter assessment post VATS surgery and subsequent Zephyr Valve insertion.
  Interventions: Procedure: Video-assisted thoracoscopic surgery (VATS) fissure completion; Device: Zephyr Valve insertion

INTERVENTIONS:
Procedure: Video-assisted thoracoscopic surgery (VATS) fissure completion — Following Bronchoscopy and Chartis® balloon catheter assessment under general anaesthesia and confirmation of collateral ventilation, a unilateral VATS lobar fissure completion will be undertaken with buttressed staples and Coseal spray intended to eliminate collateral ventilation.
Device: Zephyr Valve insertion — Following fissure completion surgery, subjects confirmed to be collateral ventilation negative will undergo bronchoscopic insertion of Zephyr® Valve(s) in the targeted lobe, under sedation or general anaesthesia.
  Other Names: Bronchoscopic Lung Volume Reduction (BLVR)

SUMMARY:
Prospective, multi-centre, pilot study aimed to evaluate the effect of Video Assisted Thoracic Surgery (VATS) fissure completion on the efficacy of endobronchial valve insertion (Zephyr Valve) in the treatment of subjects with severe Chronic Obstructive Pulmonary Disease (COPD) who exhibit collateral ventilation.

DETAILED DESCRIPTION:
The study will be a prospective, multi-centre, pilot study aimed to evaluate the effect of VATS fissure completion on the efficacy of endobronchial valve insertion (Zephyr Valve) in the treatment of subjects with severe COPD who exhibit collateral ventilation.

Study patients who provide informed consent and meet the initial inclusion/exclusion criteria following baseline screening assessments and multidisciplinary review to determine eligibility will undergo two procedures, not less than 28 days apart. The first procedure will involve an initial bronchoscopy and Chartis® assessment of collateral ventilation under general anaesthesia followed by a VATS fissure completion between targeted lobes in subjects that have collateral ventilation. The second procedure undertaken following fissure completion surgery will involve bronchoscopic insertion of Zephyr® Valve(s) in the targeted lobe, under sedation or general anaesthesia.

Subjects will be followed up over a 6-month period following VATS fissure completion and Zephyr® Endobronchial Valve (Zephyr Valve) insertion.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to provide informed consent and to participate in the study.
2. Subject is ≥ 40 years of age.
3. Subject has a diagnosis of severe or very severe homogenous or heterogeneous COPD (Global Initiative for Obstructive Lung Disease (GOLD) classification).
4. Subject has a post bronchodilator 15% ≤ FEV1 ≤ 50%.
5. Subject has Total Lung Capacity (TLC) ≥ 100% predicted.
6. Subject has Residual Volume (RV) ≥ 150% predicted.
7. Subject has a normal dobutamine stress echocardiogram.
8. Subject has sufficient exercise tolerance i.e. 150m ≤ 6MWT ≤ 450m.
9. Subject has an incomplete lobar fissure i.e. < 90%, as confirmed by CT evaluation of lung fissures.
10. Collateral ventilation confirmed as assessed by Chartis Assessment (to be confirmed during first procedure/operation)
11. Subject has stopped smoking for at least 8 weeks prior to entering the study as confirmed by carboxyhaemoglobin or cotinine levels.
12. Subject is up to date with preventive vaccinations including seasonal influenza vaccine and pneumococcal vaccine consistent with the Victorian Department of Health and Human Services Immunization Schedule Guidelines (updated March 2018).

Exclusion Criteria:

1. Subject has a history of previous thoracotomy, lung volume reduction surgery, prior lobectomy or pneumonectomy, prior lung transplantation, prior airway stent placement, prior pleurodesis, or prior endobronchial lung volume reduction therapy of any form.
2. Subject has an acute COPD exacerbation.
3. Subject has evidence of active respiratory infection.
4. Subject has a post bronchodilator FEV1 < 15%.
5. Subject has a Diffusing capacity for carbon monoxide (DLCO) < 20%.
6. Subject has a history of recurrent clinically significant respiratory infections, defined as three (3) or more COPD exacerbations requiring hospitalization during the 12 months prior to study enrollment (Informed Consent Form signature page).
7. Subject has severe gas exchange abnormalities as defined by any one of the following:

   1. Partial pressure of oxygen (PaO2) < 60 mmHg
   2. Partial pressure of carbon dioxide (PaCO2) > 45 mmHg
   3. Oxygen saturation (SpO2) < 90% on ≥ 4 L/min supplemental O2 at rest
8. Subject use of systemic steroids > 20mg/day or equivalent and/or immunosuppressive agents in the 4 weeks prior to procedure.
9. Subject unable to temporarily interrupt use of heparins or oral anticoagulants or antiplatelet agents, excluding aspirin.
10. Subject's pre-operative CT scan indicates the presence of any of the following radiological abnormalities:

    1. Pulmonary nodule ≥ 0.8 cm in diameter (does not apply if present for 2 years or more without increase in size or if proven benign by biopsy/positron emission tomography (PET)).
    2. Radiological picture consistent with active pulmonary infection, e.g. unexplained parenchymal infiltrate.
    3. Giant bullae > 30% of the volume of either lung.
    4. Significant interstitial lung disease.
    5. Significant pleural disease.
11. Subject's baseline electrocardiogram (ECG) demonstrates clinically significant arrhythmias or conduction abnormalities.
12. Clinically significant asthma (reversible airway obstruction), chronic bronchitis or bronchiectasis.
13. Subject has a known diagnosis of alpha-1 antitrypsin deficiency.
14. Subject is classified as having "likely" pulmonary hypertension defined as tricuspid regurgitation velocity > 3.4m/s and/or pulmonary artery peak systolic pressure > 45 mmHg on echocardiogram or a previous formal diagnosis of pulmonary hypertension on right heart catheterization.
15. Subject has suspected significant coronary artery disease defined as regional wall motion abnormalities on dobutamine stress echocardiogram.
16. Subject is classified as being at major cardiac risk with the presence of unstable coronary syndromes (i.e. unstable or severe angina or recent myocardial infarct), decompensated heart failure, significant arrhythmias or severe valvular disease, which warrants intensive management of the condition in accordance with current guidelines on perioperative cardiovascular risk.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Residual Volume (RV) | 6 months
  Absolute Change in Residual Volume (RV) from baseline to 6-months post Zephyr Valve procedure.

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | 6 months
  Absolute change in Forced Vital Capacity (FVC) from baseline to 6-months post Zephyr Valve procedure.
Forced Expiratory Volume in 1 second/Forced Vital Capacity (FEV1/FVC) | 6 months
  Absolute change in FEV1/FVC ratio from baseline to 6-months post Zephyr Valve procedure.
Total Lung Capacity (TLC) | 6 months
  Absolute change in Total Lung Capacity (TLC) from baseline to 6-months post Zephyr Valve procedure.
Six-Minute Walk Test (6MWT) | 6 months
  Absolute change in Six-Minute Walk Test (6MWT) from baseline to 6-months post Zephyr Valve procedure.
St. George's Respiratory Questionnaire (SGRQ) Total Score | 6 months
  Absolute change in the St. George's Respiratory Questionnaire Total Score from Baseline to 6-months post Zephyr Valve procedure. The St. George's Respiratory Questionnaire measures health status (quality of life) in patients with diseases of airways obstruction. Scores range from 0 to 100, with higher scores indicating more limitations.
Modified Medical Research Council (MMRC) Score | 6 months
  Absolute change in the modified Medical Research Council (MMRC) Score from Baseline to 6-months post Zephyr Valve procedure. The mMRC (Modified Medical Research Council) stratifies severity of dyspnea in respiratory diseases. The severity of dyspnea is rated on a scale of 0 to 4, with higher scores indicating more limitations.
Forced Expiratory Volume in 1 second (FEV1) | 6 months
  Percent change in FEV1 from baseline to 6-months post Zephyr Valve procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Alam, MD, Principal Investigator — St Vincent's Hospital Melbourne
Locations (2):
- Australia (2):
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - St. Vincent's Private Hospital Fitzroy, Fitzroy, Victoria

IPD SHARING:
Plan to Share IPD: No